CLINICAL TRIAL: NCT01635231
Title: Effect of Thiazide, Amiloride and Hypertonic Saline on Sodium- and Water Channel Activity in the Nephron in Healthy Subjects Estimated by Urinary Biomarkers
Brief Title: The Effect of Thiazide, Amiloride and Hypertonic Saline on Urinary Biomarkers in Healthy Subjects
Acronym: THAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Ph.d student Janni Majgaard Jensen, Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EBP-JMJ-2012-1
Record Dates: First submitted 2012-06-13; First posted 2012-07-09 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Nephropathy
Keywords: Nephrology; sodium-channels; water-channels; BCM; central blood pressure
MeSH Terms: conditions — Kidney Diseases | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- thiazide, diuretic (Active Comparator): 1.25 mg thiazide twice daily for 5 days
  Interventions: Other: hypertonic saline
- amiloride, diuretic (Active Comparator): 5 mg of amiloride twice daily
  Interventions: Other: hypertonic saline
- calcium (Placebo Comparator): placebo twice daily for 5 days
  Interventions: Other: hypertonic saline

INTERVENTIONS:
Other: hypertonic saline — hypertonic saline 3.0% 7 ml/kg
  Other Names: NaCl 3.0 %

SUMMARY:
Urinary biomarkers (u-NKCC2, u-ENaC-gamma and u-AQP2) reflects the activity of the sodium- and water channels in the human kidney.

Changes in the sodium-and water channel activity can be induced by blocking the sodium channels with diuretics in healthy subjects

DETAILED DESCRIPTION:
1. Urinary biomarkers (u-NKCC2, u-ENaC-gamma and u-AQP2) reflects the kidneys transport of sodium and water in the nephron.
2. Changes in the sodium-and water channel activity is induced by blocking the NCC channels with thiazide and ENaC channels with amiloride and by intervention with hypertonic NaCl The changes in sodium-and water channels are followed by changes in extracellular and intracellular fluids, central bloodpressure and the plasma concentration of vasoactive hormones.

The purpose of this study is to investigate the changes in urinary biomarkers (u-NKCC2, u-ENaC-gamma and u-AQP2), extra- and intracellular fluid compartments, central bloodpressure and the plasma concentration of Vasoactive hormones in healthy subjects under a) treatment with Amiloride and Thiazide at baseline and b) after and acute infusion with hypertonic saline.

Subjects will be examined on three examination days. Four days prior to the examination days the subjects will consume a standard diet based on amount of sodium and calories and randomized to treatment with either thiazide, amiloride or placebo twice daily for 5 days. On the examination days the subjects receive an infusion with hypertonic saline.

Renal function is measured by renal clearance of 51Cr-EDTA. Urinary biomarkers (u-NKCC2, u-ENaC-gamma and u-AQP2) will be measured to evaluate the activity of water- and sodium channels in the nephron, changes in fluid compartments are measured by body composition monitor. Central blood pressure is measured by sphygmocor.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females
* age 18-45
* BMI range 18,5-30,0 kg/m2

Exclusion Criteria:

* hypertension (i.e. ambulatory BP > 130 mmHg systolic or/and > 80 mmHg diastolic)
* history or clinical significant signs of heart, lung, liver, kidney, endocrine, brain or neoplastic
* disease.
* alcohol abuse
* drug abuse
* smoking
* pregnancy or nursing
* blood donation within a month prior to examination
* medical treatment apart from oral contraception abnormal blood samples, -ECG and -urine dipstick, drug abuse, alcohol abuse, pregnancy, medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
urinary biomarkers | baseline, 0 hours and 1.5 hours after intervention
  Urinary excretion of epithelial sodium channels (ENaC), Sodium-potassium-2chloride transporters (NKCC2) and aquaporin2 channels (AQP2) before, during and after fluid infusion

SECONDARY OUTCOMES:
vaso active hormones | baseline, 0 hours and 1.5 hours after intervention
  plasma concentrations of: renin, Angiotensin II, aldosterone, Vasopressin, ANP and BNP
central blood pressure | baseline, 0 hours and 1.5 hours after intervention
  measured by applanation-tonometry
intracellular (ICV)- and extracellular volume (ECV) | baseline, 0 hours and 1.5 hours after intervention
  change in ICV and EVC from baseline and after intervention measured in liters by body composition monitor (BCM)

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, MD, DMSc, Study Director — Medical Research, Holstebro
Locations (1):
- Medical Research, Holstebro, Denmark